CLINICAL TRIAL: NCT02077127
Title: Association of Monocyte Chemoattractant Protein-1 (MCP-1)2518A/G Polymorphism With Proliferative Diabetic Retinopathy in Northern Chinese Type 2 Diabetes
Brief Title: Monocyte Chemoattractant Protein-1 2518A/G Polymorphism
Acronym: MCP-1
Status: Completed | Type: Observational
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Li Dong, Li Dong, Harbin Medical University
Other Study IDs: dongli
Record Dates: First submitted 2013-06-10; First posted 2014-03-04 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood had been stored in -80℃.
Oversight: Data Monitoring Committee: No

SUMMARY:
The pathogenesis of proliferative diabetic retinopathy (PDR) remains poorly understood. Recent studies have implicated that monocyte chemoattractant protein-1 (MCP-1) is associated with diabetic microvascular or macrovascular complications. However, the relationship between SNP polymorphism c.2518A/G in the MCP-1 gene with diabetic retinopathy remains controversial. In the present study, we evaluated the association of a single nucleotide polymorphism (SNP) in the MCP-1 gene with diabetic retinopathy (DR) and diabetic macular edema (DME) in Chinese population from Southern China with type 2 diabetes.

DETAILED DESCRIPTION:
The association between polymorphism of MCP-1 c.2518A/G and DR had been reported in Japan and Korea, but their opinion were inconsistent. However there is no report in China so far. This study was designed to clarify the relationship of polymorphism of MCP-1 c.2518A/G with type 2 diabetes with or without DR. The relationship between MCP-1 c.2518A/G and different stage of DR has also been studied.This article proved that the MCP-1 c.2518G/G genotype is a susceptibility gene for DR in Chinese type 2 diabetic patients, especially the High-risk PDR. There is no association with DME and c.2518G/G.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic retinopathy
* age at diagnosis ≥30 years and a known duration of diabetes of ≥5 years.

Exclusion Criteria:

* eyeball atrophy
* epimacular membrane
* age-related macular degeneration (ARMD)
* intravitreal injection medicine
* vitreous hemorrhage

Ages: 41 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: residents of a certain province
Sampling Method: Non-Probability Sample
Enrollment: 1043 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Genetic association | 1 year
  age at diagnosis of diabetes ≥30 years and a known duration of diabetes of ≥5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liu, Doctor, Study Chair — First Affiliated Hospital of Harbin Medical University
Locations (1):
- Harbin Medical University, Harbin, Heilongjiang, China